CLINICAL TRIAL: NCT07168343
Title: The Effect of Two Icodextrin Exchanges on Fluid Status and Blood Pressure Control in Children on Chronic Peritoneal Dialysis
Brief Title: Effectiveness of Two Icodextrin Exchanges on Fluid Status and Blood Pressure Control Compared to a Single Icodextrin Exchange
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National University Health System, Singapore (Other)
Collaborators: The UCL Great Ormond Street Institute of Child Health (Other); Children's Hospital of Fudan University (Other); Philippine Children's Medical Center (Other Government)
Responsible Party: Principal Investigator, Sharon Teo, Consultant, National University Health System, Singapore
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2024-4140
Record Dates: First submitted 2025-09-04; First posted 2025-09-11 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Children on Chronic Peritoneal Dialysis
Keywords: Children; CAPD; CCPD; Icodextrin

STUDY DESIGN:
Intervention Model Description: Total study duration is 12 weeks. 4-week run-in period 4 weeks in one icodextrin exchange 4 weeks in two icodextrin exchanges according to randomization. There will be 3 study visits at baseline, 4 and 8 weeks.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (1-Ico) (Active Comparator): Group A (One icodextrin exchange followed by two icodextrin exchanges)
  Interventions: Drug: One icodextrin exchange; Drug: Two icodextrin exchanges
- Group B (2-Ico) (Experimental): Group B (Two icodextrin exchanges followed by one icodextrin exchange)
  Interventions: Drug: One icodextrin exchange; Drug: Two icodextrin exchanges

INTERVENTIONS:
Drug: One icodextrin exchange — One icodextrin fill volume of 550ml/m2 body surface area which is optimal for most paediatric patients is recommended. The minimum dwell time for an icodextrin exchange will be 7 hours, and range between 7-10 hours.
  Other Names: 1-Ico
Drug: Two icodextrin exchanges — In two icodextin exchanges, the dwell times can vary but must be a minimum of 7 hours.
  Other Names: 2-Ico

SUMMARY:
Fluid overload and hypertension are prevalent in children undergoing chronic peritoneal dialysis (PD), especially in low- and middle-income countries (LMICs). These complications often lead to increased hospitalizations, higher medication use, and, in some cases, conversion to hemodialysis. Icodextrin is used to enhance ultrafiltration (UF) and reduce glucose exposure, but its effectiveness in children with a single long dwell has been inconsistent. Preliminary observations suggest that shorter, twice-daily icodextrin exchanges may improve UF and blood pressure (BP) control. However, no randomized trial has evaluated this approach in pediatric patients.

DETAILED DESCRIPTION:
1. Background and Rationale Fluid overload and hypertension are among the most prevalent and clinically significant complications in pediatric patients receiving chronic peritoneal dialysis (PD). In children, extracellular volume expansion contributes to left ventricular hypertrophy, increased arterial stiffness, impaired growth, and heightened cardiovascular morbidity and mortality. These complications are especially burdensome in low- and middle-income countries (LMICs), where limited access to automated PD, hemodialysis facilities, and antihypertensive medications leads to frequent hospitalizations, increased costs, and higher rates of dialysis modality switch.

   Icodextrin is a glucose polymer solution used in PD as a glucose-sparing osmotic agent. Unlike glucose-based solutions that rely on crystalloid osmosis and are subject to rapid dissipation of the osmotic gradient, icodextrin provides sustained ultrafiltration (UF) through colloid osmosis. Its absorption via lymphatic pathways leads to more stable osmotic gradients, particularly during long dwell periods. However, pediatric studies show inconsistent results when icodextrin is used once daily in a single long daytime dwell, with some children demonstrating inadequate fluid removal and variable blood pressure (BP) control.

   Emerging observational data and small pilot studies suggest that dividing the icodextrin dose into two separate exchanges per day (2-Ico) may improve ultrafiltration efficiency by maintaining a more consistent osmotic gradient throughout the 24-hour cycle. This approach may also reduce fluctuations in intravascular volume, improve BP stability, and enhance patient comfort. To date, however, no randomized controlled trial (RCT) has rigorously assessed the safety, efficacy, and tolerability of two daily icodextrin exchanges in the pediatric population.

   This investigator-led multicenter randomized crossover trial addresses this evidence gap and aims to determine whether two daily icodextrin exchanges improve fluid status, BP control, and patient-related outcomes compared with a single daily icodextrin exchange in children on chronic PD.
2. Study Objectives

Primary Objective:

• To determine whether two daily icodextrin exchanges (2-Ico) provide superior ultrafiltration and blood pressure control compared to one daily icodextrin exchange (1-Ico) in children on PD.

Secondary Objectives:

* To evaluate the effect of 2-Ico versus 1-Ico on:

  1. Objective measures of fluid status (bioimpedance spectroscopy, interdialytic weight change, ambulatory BP monitoring).
  2. Solute clearance parameters, including Kt/V and creatinine clearance.
  3. Safety and tolerability, including infection rates, biochemical complications, and episodes of symptomatic hypotension.
  4. Patient- and caregiver-reported quality-of-life outcomes, treatment satisfaction, and burden of care.

  3. Study Hypothesis Two daily icodextrin exchanges are safe, feasible, and more effective than a single daily exchange in improving fluid overload and BP control in children receiving chronic PD.

  4. Study Design This is a prospective, multicenter, randomized, open-label, crossover trial.
* Population (P): Children aged 5-18 years on CAPD or CCPD for ≥4 weeks with persistent hypertension (mean arterial pressure >95th percentile on 24-hour ABPM or requiring antihypertensive medication).
* Intervention (I): Two icodextrin exchanges per day (2-Ico).
* Comparator (C): One icodextrin exchange per day (1-Ico).
* Outcomes (O): Primary - change in 24-hour ultrafiltration volume. Secondary - changes in fluid status, BP, solute clearance, safety, and patient-reported outcomes.
* Timeframe (T): 12-week participation per patient, including a 4-week run-in and two 4-week randomized intervention phases (crossover design).

Randomization and Crossover:

Participants will be randomized 1:1 to either sequence (1-Ico → 2-Ico or 2-Ico → 1-Ico) following the run-in period. No washout is required, as each phase is of sufficient duration to reflect steady-state physiology.

5. Intervention Details

Icodextrin Prescription:

* Fill volume: 550 mL/m² body surface area (BSA), based on pediatric optimization studies (Rousso et al., Pediatr Nephrol 2016; doi:10.1007/s00467-016-3398-1).
* Minimum dwell time: 7 hours (acceptable range 7-10 hours).
* Total daily exposure: one or two exchanges depending on allocation arm.

CAPD Program:

* Standard CAPD: four daily exchanges.
* 1-Ico arm: One icodextrin dwell (typically overnight), with three glucose-based dwells.
* 2-Ico arm: Two icodextrin dwells (overnight and first daytime dwell), with two glucose-based dwells.
* To minimize cost, one icodextrin bag may be aseptically split for two exchanges without patient disconnection. Families will receive structured retraining to reduce infection risk.

CCPD Program:

* Standard CCPD: nocturnal automated glucose-based exchanges followed by a long daytime dwell.
* 1-Ico arm: One icodextrin dwell (daytime).
* 2-Ico arm: Two icodextrin dwells (one daytime, one post-school dwell, each ≥7 hours).

Adjunct Management:

* Glucose-based PD fluid strength and dwell times may be adjusted by treating physicians according to patient volume status.
* Fluid and sodium intake restrictions will remain constant throughout the study.
* All changes will be recorded on standardized case report forms. 6. Outcomes

Primary Outcome:

• Mean change in 24-hour ultrafiltration volume between 1-Ico and 2-Ico phases.

Secondary Outcomes:

1. Fluid Status:

   1. Bioimpedance spectroscopy (extracellular water/total body water ratio).
   2. Interdialytic weight change.
   3. Ambulatory BP monitoring (24-hour mean, systolic/diastolic load).
2. Solute Clearance:

   1. Weekly Kt/V (urea).
   2. Creatinine clearance (mL/min/1.73m²).
3. Safety and Tolerability:

   1. Incidence of peritonitis and exit-site infections.
   2. Symptomatic hypotension episodes.
   3. Electrolyte disturbances (hyponatremia, hypokalemia).
   4. Biochemical safety parameters (glucose, serum lipids).
4. Patient- and Caregiver-Reported Outcomes:

   1. Quality of life (PedsQL questionnaire).
   2. Treatment satisfaction (Likert scale surveys).
   3. Caregiver burden (validated caregiver strain index).

7. Risks and Benefits

Risks:

* Physical: venipuncture discomfort, transient hypotension, peritonitis due to additional bag handling.
* Psychological: survey-related stress, inconvenience of post-school exchange.
* Data: low risk of confidentiality breach (mitigated by secure data management).

Benefits:

* Direct: Improved fluid control, BP stabilization, and potential reduction in hospitalizations and antihypertensive medication use.
* Indirect: Evidence generation to guide PD practice in LMICs, increased global knowledge on icodextrin optimization in pediatric PD.

ELIGIBILITY:
Inclusion Criteria:

1. Children 5-18 years of age
2. Receiving CAPD or CCPD for at least the preceding 4 weeks, and not likely to change from CAPD to CCPD during the study period
3. 24-hour mean arterial pressure (MAP; measured by ambulatory blood pressure monitoring (ABPM) above the 95th percentile for age, sex, and height
4. 24-hour urine output less than 200ml/day

Exclusion Criteria:

1. Children under 5 years of age (as younger children are more prone to hyponatremia)
2. Children with systolic BP < 50th centile for age, sex, and height in the preceding 4 weeks)
3. Children who are polyuric or those prone to hypotension (defined as > 2 episodes of systolic BP < 5th centile in the 4 weeks preceding the study)
4. Known allergy to starch
5. Pregnant women
6. Patients with maltose or isomaltose intolerance, glycogen storage disease, pre-existing severe lactic acidosis, uncorrectable mechanical defects that prevent effective PD or increase the risk of infection and documented loss of peritoneal function or extensive adhesions that compromise peritoneal function

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Estimated)
Dates: Start 2026-02-28 (Estimated); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Ultrafiltration efficiency | 12 weeks
  Ultrafiltration (UF): Assessed clinically through blood pressure, presence of edema or crackles, reduced need for antihypertensive medications, residual kidney function, and mean daily UF.
The solute clearance adequacy | 12 weeks
  Toxin Removal: Evaluated by comparing pre- and post-intervention levels of electrolytes and urea clearance, calculated using the Kt/V formula.

SECONDARY OUTCOMES:
To measure caregiver burden | 12 weeks
  Caregiver burden will be measured by using a Paediatric Renal Caregiver Burden Scale (PR-CBS) Using the Caregiver Burden Scale (1-5, with higher scores indicating greater burden), we will assess whether the additional exchange is perceived as an increased burden or a relief, particularly if clinical improvements in the child are observed.

CONTACTS AND LOCATIONS:
Locations (1):
- National University Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No
Only de-identified data will be shared.